CLINICAL TRIAL: NCT05189431
Title: Predictive Power of Peripheral Perfusion Index During Induction of Aneasthesia
Brief Title: Peripheral Perfusion Index During Induction of Anaesthesia
Status: Completed | Type: Observational
Sponsor: Jakob Højlund (Other)
Responsible Party: Sponsor-Investigator, Jakob Højlund, Assistant professor, consultant, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: H-19016524
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia
Keywords: monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We wish to study the feasibilty of using the peripheral perfusion index as a supplementary monitor during induction of general anesthesia

DETAILED DESCRIPTION:
Haemodynamic monitoring during general anaesthesia (GA) traditionally relies on simple and readily available parameters such as blood pressure and heart rate. Most patients will only have intermittent non-invasive monitoring of blood pressure. During the induction phase an abrupt reduction in blood pressure is often seen, with possible deleterious consequences for organ perfusion [1,2]. The availability of continuous monitoring of systemic haemodynamics is limited by cost and scarcity of equipment and personnel.

The peripheral perfusion index (PPI) is obtained non-invasively by photoplethysmography - ubiquitously present in the perioperative setting [3,4]. The PPI is a simple ratio describing the proportion of pulsatile to non-pulsatile signal attenuation. No specialized equipment is needed as the PPI is inherent to photoplethysmography already ubiquitous during GA, although not all pulse-oxymeters are set up to display PPI. The PPI in awake patients is dominated by sympathetic tone [4] creating a highly positively skewed distribution [3]. Conversely, during GA cardiac stroke volume (SV) becomes the major determinant of PPI [5,6]. Very little evidence exists regarding the efficacy of PPI as a monitor during the induction of GA. Presumably, the net effect will be a composite of two opposing mechanisms: Sympatholysis increasing PPI, with decreased SV/CO causing the opposite effect.

The present study was designed to explore the clinical utility of the non-invasively obtained peripheral perfusion index to detect cardiovascular compromise during induction of general anaesthesia. We hypothesized that during induction of GA changes in systemic haemodynamics in the form of mean arterial pressure (MAP) and cardiac stroke volume (SV) and -output (CO) during GA would be reflected in the PPI, albeit in a complex manner. Thus, a predominant vasodilatory response might be differentiated from a response dominated by decreased CO.

1. Sessler DI, Meyhoff CS, Zimmerman NM, Mao G, Leslie K, Vásquez SM, et al. Period-dependent Associations between Hypotension during and for Four Days after Noncardiac Surgery and a Composite of Myocardial Infarction and Death. Anesthesiology [Internet]. 2018 [cited 2018 Nov 30];128:317-27. Available from: http://www.ncbi.nlm.nih.gov/pubmed/29189290
2. Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, et al. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery. Anesthesiology [Internet]. 2017 [cited 2018 Nov 30];126:47-65. Available from: http://www.ncbi.nlm.nih.gov/pubmed/27792044
3. Lima AP, Beelen P, Bakker J. Use of a peripheral perfusion index derived from the pulse oximetry signal as a noninvasive indicator of perfusion. Crit Care Med [Internet]. 2002 [cited 2018 Jan 11];30:1210-3. Available from: http://www.ncbi.nlm.nih.gov/pubmed/12072670
4. Reisner A, Shaltis PA, McCombie D, Asada HH. Utility of the photoplethysmogram in circulatory monitoring. Anesthesiology. 2008;108:950-8.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery under general anesthesia

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of general populace for surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in systemic hemodynamics at 2 minutes | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Højlund, MD, Principal Investigator — Dept. Anesthesiology, Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital Region, Denmark

DOCUMENTS (1):
  • Study Protocol (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05189431/Prot_000.pdf